CLINICAL TRIAL: NCT03865862
Title: Efficacy of Load Control in Eccentric Exercises in the Increase of the Cross-sectional Area and Pain Threshold of the Patellar Tendon, and of the Strength of the Quadriceps in Volleyball Players. A Randomized Clinical Trial
Brief Title: Load Control in Eccentric Exercises in Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEX
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Patellar Abnormality
Keywords: Eccentric; Load control; Volleyball; Physiotherapy; Patellar tendon; Randomized clinical trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Intervention of 4 weeks, with two weekly sessions, in which the intervention will be carried out during the training, these sessions having a duration of 10 minutes. During the performance of the intervention, they will perform 3 sets of 15 repetitions of squats in a 25º inclined plane, performing the eccentric phase of the squat in a time of 4 seconds, the concentric phase in 3 seconds, and a rest of 15 seconds between series.
  Interventions: Other: Experimental
- Control (Active Comparator): Intervention of 4 weeks, with two weekly sessions, in which the intervention will be carried out during the training, these sessions having a duration of 10 minutes. During the performance of the intervention, they will perform 3 sets of 15 repetitions of squats in a 25º inclined plane, performing the eccentric phase of the squat in a time of 4 seconds, the concentric phase in 3 seconds, and a rest of 15 seconds between series.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The athletes will perform an intervention of 4 weeks, with two weekly sessions, in which the intervention will be performed during the training, with these sessions lasting 10 minutes. During the performance of the intervention, they will perform 3 sets of 15 repetitions of squats in a 25º inclined plane, performing the eccentric phase of the squat in a time of 4 seconds, the concentric phase in 3 seconds, and a rest of 15 seconds between series. This intervention will be performed adding 50% of his OR as external load during the first two weeks, 55% of his MR during the third week, and 60% of his MR in the fourth week of the intervention. During the exercise you can help the physiotherapist who will accompany you to perform the concentric phase without load.
  Other Names: Load control in eccentric exercises
  Arms: Experimental
Other: Control — Intervention of 4 weeks, with two weekly sessions, in which the intervention will be carried out during the training, these sessions having a duration of 10 minutes. During the performance of the intervention, they will perform 3 sets of 15 squat repetitions on a 25º inclined plane, performing the eccentric phase of the squat in a time of 4 seconds, the concentric phase in 3 seconds, and a 15-second rest between series. The subjects of this group will perform the protocol using only their own weight as a load.
  Other Names: Eccentric exercises
  Arms: Control

SUMMARY:
Introduction. Vertical jump is the main movement in volleyball, and the main etiological factor of patellar tendinopathy. The eccentric exercise has been proved as the most effective intervention in improving this factor.

Aim. Annalise the effectiveness of the load control during the eccentric exercise to increase the cross-sectional area as well as the increase of the pain threshold of the patellar tendon, and the gain of the quadriceps maximum strength, in volleyball older players.

Study design. Randomized clinical study, simple blind, multicentric and with a follow-up period.

Methods. 40 volleyball players will be recruited, who will be randomized to the two groups: experimental (control of the load based on the RM during the eccentric exercise of quadriceps) and control (without load control). There will be an intervention of 4 weeks with 2 weekly seasons of 10 minutes each. The dependent variables will be: cross-sectional area (ultrasound evaluation), pain threshold in the patellar tendon (analog or digital algometer) and the maximum strength of the quadriceps (linear encoder or estimating the RM). In case of normality of the distribution of the sample, parametric tests will be used: student t-test of related samples (difference between evaluations in each rump) and repeated measures ANOVA (intra- and intergroup effect).

Expected results. To observe an increase in the cross-sectional area, pain-threshold of patellar tendon and quadriceps maximum strength.

ELIGIBILITY:
Inclusion Criteria:

* Volleyball players
* Federated that at the time of the study compete in clubs of the Community of Madrid
* Over 18 years old.

Exclusion Criteria:

* Present a medical diagnosis of injury or illness
* Have suffered a knee injury in the 6 months prior to the study
* Doing some pharmacological or physiotherapy treatment external to the study
* Not signed the informed consent document.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline cross-sectional area of the patellar tendon after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the cross-sectional area of the patellar tendon will be assessed by ultrasound measurement. The player must be in the supine position, with the lower limbs resting on a wedge while maintaining a knee flexion of 15-20º. The physiotherapist will make a measurement with the transversal axis of the ultrasound, 1 cm distal to the lower pole of the patella, and with the longitudinal axis to 0.5cm distal of the same pole. In spite of performing the measurement of both lower limbs, only the data of the cross-sectional area of the patellar tendon of the dominant lower limb used by the athlete during the landing of the jump while playing will be analyzed. The unit of measurement will be the centimeter. A higher score in the post-treatment evaluation indicates an improvement in the cross-sectional area of the patellar tendon.

SECONDARY OUTCOMES:
Change from baseline pain threshold to pressure after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the pain threshold to the pressure of the patellar tendon will be quantified using a digital algometer. During the measurement, the subject will remain in the supine position, maintaining a knee flexion of 15-20º supported by a wedge. The physiotherapist will apply the algometer directly on the lower edge of the patella, towards the proximal side of the tendon. As in the previous test, despite evaluating the pressure threshold in both lower limbs, only the result of the dominant lower limb will be counted. This test is quantified on a 0-100 points scale, where a higher score will indicate a greater perception of pain under pressure.
Change from baseline maximum strength of quadriceps after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the maximum strength of quadriceps will be an estimate of the MRI, where the subjects, after warming up, will begin the test by raising a load estimated by themselves of their 80% MR and will progressively increase the load to 1 repetition (if the repetition is correct will continue to gain weight until the failed attempt). They will have 5 total attempts resting 1 minute between each attempt. The unit of measurement is the Kg, where a greater amount indicates a greater maximum strength of quadriceps.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain